CLINICAL TRIAL: NCT00537004
Title: Asymmetric Neurodegeneration and Language in Primary Progressive Aphasia
Brief Title: Language in Primary Progressive Aphasia
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Marsel Mesulam, Director, Mesulam Center for Cognitive Neurology and Alzheimer's Disease, Northwestern University
Other Study IDs: IA0125; R01AG077444 (NIH)
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Primary Progressive Aphasia
Keywords: primary progressive aphasia; frontotemporal dementia; semantic dementia; progressive nonfluent aphasia; progressive aphasia; frontotemporal lobar degeneration
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia; Primary Progressive Nonfluent Aphasia; Aphasia; Frontotemporal Lobar Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PPA (Primary Progressive Aphasia): Individuals with primary progressive aphasia
- Control: Individuals with no diagnosis of any type of dementia

SUMMARY:
The purpose of this study is to further define the neurological and linguistic deterioration in primary progressive aphasia.

DETAILED DESCRIPTION:
The Language in Primary Progressive Aphasia (PPA) aims to understand the behavioral, anatomical and physiological changes in people with PPA throughout the course of the illness. The researchers in this study want to increase awareness of PPA, educate others about this unique disorder, and to encourage more research to eventually develop therapies.

During the three-day research program, participants will be asked to undergo neuropsychological testing (paper and pencil tests that evaluate cognition), advanced imaging (MRI and PET), cognitive experiments, and other computer and language testing batteries. Participants may be asked to return every two years to complete the same measures.

For participants not living near Chicago, IL, flights and accommodations (for both the person with PPA and their companion) will be covered by the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary progressive aphasia
* Right-handed
* Native English speaker
* Visual acuity of 20/30 corrected
* Adequate hearing to follow conversation
* Safe for an MRI scan

Exclusion Criteria:

* Left-handedness
* Claustrophobia
* Presence of significant medical illness that initially or in the future could interfere with continued participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with PPA will be recruited from the Northwestern University Alzheimer's Disease Center Core registry, the Northwestern University Neurobehavior and Memory Clinic, and from those who contact the center that are interested in PPA research.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-05 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological variables | Immediately after testing and at two years post-testing

CONTACTS AND LOCATIONS:
Overall Officials: Marsel Mesulam, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Mesulam MM. Slowly progressive aphasia without generalized dementia. Ann Neurol. 1982 Jun;11(6):592-8. doi: 10.1002/ana.410110607. PMID 7114808
- [Background] Weintraub S, Rubin NP, Mesulam MM. Primary progressive aphasia. Longitudinal course, neuropsychological profile, and language features. Arch Neurol. 1990 Dec;47(12):1329-35. doi: 10.1001/archneur.1990.00530120075013. PMID 2252450
- [Derived] Mesulam MM, Coventry C, Kuang A, Bigio EH, Mao Q, Flanagan ME, Gefen T, Sridhar J, Geula C, Zhang H, Weintraub S, Rogalski EJ. Memory Resilience in Alzheimer Disease With Primary Progressive Aphasia. Neurology. 2021 Feb 9;96(6):e916-e925. doi: 10.1212/WNL.0000000000011397. Epub 2021 Jan 13. PMID 33441454
- See also: PPA Research at Northwestern University — https://www.brain.northwestern.edu/join/index.html